CLINICAL TRIAL: NCT04933123
Title: Clinical Evaluation of a New Dental Glass Ceramic in the Indirect Restorative Therapy
Brief Title: Clinical Evaluation of a Dental Glass Ceramic
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: insufficient clinical performance which might have led to AE
Sponsor: Ivoclar Vivadent AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LL3965040
Record Dates: First submitted 2021-06-14; First posted 2021-06-21 (Actual); Results first posted 2025-04-02 (Actual); Last update posted 2025-04-20 (Actual); Status verified 2025-04

CONDITIONS: Caries; Dental Trauma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Inlay/Onlay (Experimental): shades A1, A2 and A3
  Interventions: Device: indirect restorative treatment with a glass ceramic

INTERVENTIONS:
Device: indirect restorative treatment with a glass ceramic — Inlays and onlays of glass ceramic for molars and premolars are adhesively luted.

SUMMARY:
A clinical trial with an experimental glass ceramic (shades A1, A2 and A3) to ensure the safety and efficacy of the product. It is a study with single-arm in which inlays and onlays for molars and premolars are adhesively luted.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-65 years
* Indication for indirect restorations (inlay, onlay) in molar or premolar - replacement of insufficient fillings (e.g. due to caries at margins, filling fracture, fracture of the tooth, poor quality of the surface, leaking margin, etc.) or extensive primary caries
* The occlusal area of the restoration must cover at least 1/3 of the occlusal area of the tooth.
* Participant wishes a restoration within the scope of the study (signed informed consent after detailed explanation and study of the patient information)
* Pre-operative discomfort of the tooth to be restored should not exceed 3 on the visual analogue scale (VAS) (0=no pain, 10=maximum conceivable pain) due to temperature stimulus or bite sensitivity
* Max. 2 restorations per participant in different quadrants.
* Healthy periodontium, no active periodontitis
* Contact with adjacent teeth (at least at one side) and opposing teeth present with at least one contact point.
* Sufficient language skills

Exclusion Criteria:

* Sufficient isolation not possible, dry working field cannot be guaranteed
* Participants with a proven allergy to one of the ingredients of the materials used
* Participants with proven allergy to local anaesthetics
* High caries activity/ poor oral hygiene
* Participants with severe systemic diseases
* Pregnancy
* Symptoms of SARS (severe acute respiratory syndrome)-CoV2 (Corona Virus 2) infection

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2021-09-14 (Actual); Primary Completion 2021-11-15 (Actual); Study Completion 2021-11-15 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Ivoclar Vivadent, Schaan, Liechtenstein

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The recruitment period lasted from 14.09.2021-15.11.2021 in the dental clinic.
Units Other Than Participants: Inlays/Onlays
Period: Overall Study
Arm/Group | Inlay/Onlay
Started | 13; 13 Inlays/Onlays
Completed | 13; 13 Inlays/Onlays
Not Completed | 0; 0 Inlays/Onlays

BASELINE CHARACTERISTICS:
Arm/Group | Inlay/Onlay
Number analyzed (Participants) | 13
Age, Customized [Number; unit: participants]
  18-65 years old | 13
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 11
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Survival Rate of Inlays and Onlays
Description: Inlay and onlay restorations were examined by a dentist
Time Frame: Baseline (7-10 days after insertion of restoration)
Measure: Number; unit: Inlays/Onlays
Units Other Than Participants: Inlays/Onlays
Arm/Group | Inlay/Onlay
Number analyzed (Participants) | 13
Number analyzed (Inlays/Onlays) | 13
Inlays/Onlays | 13

2. Secondary Outcome: Quality Criteria (Modified FDI Criteria)
Description: assessed following the FDI criteria on a scale from 1 "very good" to 5 "unacceptable" (e.g. surface lustre, Staining, fracture of material, retension, occlusal contour and wear, and colour match of restorations)
Time Frame: Baseline (7-10 days after insertion of restoration)
Measure: Number; unit: inlays/onlays
Units Other Than Participants: Inlays/Onlays
Arm/Group | Inlay/Onlay
Number analyzed (Participants) | 13
Number analyzed (Inlays/Onlays) | 13
inlays/onlays
  FDI 1 (Surface Luster), FDI Score 1 | 13
  FDI 1 (Surface Luster), FDI Score 2-5 | 0
  FDI 2a (Surface Staining), FDI Score 1 | 13
  FDI 2a (Surface Staining), FDI Score 2-5 | 0
  FDI 2b (Margin Staining), FDI Score 1 | 13
  FDI 2b (Margin Staining), FDI Score 2-5 | 0
  FDI 3 (Color Match), FDI Score 1 | 10
  FDI 3 (Color Match), FDI Score 2 | 3
  FDI 3 (Color Match), FDI Score 3-5 | 0
  FDI 3 (Translucency), FDI Score 1 | 12
  FDI 3 (Translucency), FDI Score 2 | 1
  FDI 3 (Translucency), FDI Score 3-5 | 0
  FDI 5 (Fractures of material and retention), FDI Score 1 | 8
  FDI 5 (Fractures of material and retention), FDI Score 2 | 5
  FDI 5 (Fractures of material and retention), FDI Score 3-5 | 0
  FDI 6 (Marginal adaptation), FDI Score 1 | 13
  FDI 6 (Marginal adaptation), FDI Score 2-5 | 0
  FDI 7a (Occlusal contour and wear, qualitatively), FDI Score 1 | 13
  FDI 7a (Occlusal contour and wear, qualitatively), FDI Score 2-5 | 0
  FDI 10 (Patient's view), FDI Score 1 | 13
  FDI 10 (Patient's view), FDI Score 2-5 | 0
  FDI 11 (Postoperative (hyper-)sensitivity and tooth vitality), FDI Score 1 | 12
  FDI 11 (Postoperative (hyper-)sensitivity and tooth vitality), FDI Score 2-5 | 0
  FDI 12 (Recurrence of caries (CAR), erosion, abfraction), FDI Score 1 | 13
  FDI 12 (Recurrence of caries (CAR), erosion, abfraction), FDI Score 2-5 | 0
  FDI 13 (Tooth integrity (enamel cracks, tooth fractures), FDI Score 1 | 13
  FDI 13 (Tooth integrity (enamel cracks, tooth fractures), FDI Score 2-5 | 0
  FDI 15 (Adjacent mucosa), FDI Score 1 | 13
  FDI 15 (Adjacent mucosa), FDI Score 2-5 | 0

ADVERSE EVENTS:
Time Frame: Baseline
Arm/Group | Inlay/Onlay
All-Cause Mortality (participants affected / at risk) | 0/13
Serious Adverse Events (participants affected / at risk) | 0/13
Other Adverse Events (participants affected / at risk) | 0/13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-09-07): https://cdn.clinicaltrials.gov/large-docs/23/NCT04933123/Prot_SAP_000.pdf